CLINICAL TRIAL: NCT00746785
Title: A New Pharmacotherapy for Alcohol Dependence: Olanzapine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Mind Research Network (Other)
Responsible Party: Principal Investigator, Kent Hutchison, Ph.D., Chief Science Officer, The Mind Research Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5R01AA014886 (NIH)
Record Dates: First submitted 2008-09-02; First posted 2008-09-04 (Estimated); Results first posted 2014-03-20 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-01

CONDITIONS: Alcohol Dependence
Keywords: Olanzapine
MeSH Terms: conditions — Alcoholism | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2.5 mg Olanzapine (Experimental): 2.5 mg Olanzapine
  1x per day for 12 weeks.
  Interventions: Drug: 2.5 mg Olanzapine
- 5mg Olanzapine (Active Comparator): 5 mg Olanzapine
  1x per day for 12 weeks.
  Interventions: Drug: 5mg Olanzapine
- Placebo (Placebo Comparator): Placebo
  1x per day for 12 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 2.5 mg Olanzapine — 2.5 mg
  Arms: 2.5 mg Olanzapine
Drug: 5mg Olanzapine — 5 mg
  Arms: 5mg Olanzapine
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
Craving for alcohol has been related to loss of control drinking and is a major target of biological and behavioral interventions for alcohol dependence. Our previous research has demonstrated that olanzapine (a dopamine antagonist) attenuates craving for alcohol, that a variant in the gene that expresses D4 receptors influences craving for alcohol, and that olanzapine is particularly effective at reducing craving among individuals with this variant. Pilot data from a recent 12 week trial of olanzapine indicates that olanzapine is well tolerated and that olanzapine reduces drinking, particularly among individuals with the aforementioned genetic variant. The objective of the present application is to examine the effectiveness of olanzapine (5 mg/day), as compared to olanzapine (2.5 mg/day) and a placebo control, in terms of reducing craving and alcohol use behavior among treatment seeking alcoholics. Furthermore, the present application will examine whether the effects of olanzapine on drinking outcomes are mediated by its effects on a specific putative mechanism (i.e., cue-elicited craving for alcohol) and determine whether the DRD4 VNTR polymorphism is a marker for the effectiveness of olanzapine. To that end, 202 alcohol dependent subjects will be randomly assigned to medication group and receive 12 weeks of medication. Subjects will complete follow-up assessments at 3 and 6 months after the end of the treatment. It is expected that olanzapine will significantly reduce cue-elicited craving and alcohol use behavior in a dose dependent fashion over the course of the 12 week trial and follow-up period, as compared to the placebo condition. Furthermore, it is expected that the effects of olanzapine on alcohol use behavior will be mediated by the effect of olanzapine on cue-elicited craving and that the effects of olanzapine on cue-elicited craving and alcohol use behavior will be moderated by the DRD4 VNTR, such that olanzapine will be more effective among individuals with the 7 repeat allele. The successful completion of the proposed research is expected to advance a new medication for alcohol dependence and advance genetic markers that predict the effectiveness of this medication.

DETAILED DESCRIPTION:
The first goal of the study is to determine whether olanzapine is effective at reducing cue-elicited craving (i.e., subjective craving as well as activation of the midbrain and prefrontal cortex after exposure to alcohol cues) for alcohol and reducing alcohol use in a sample of alcohol dependent subjects. The second goal is to test the putative mechanism of change by determining whether the effect of olanzapine on alcohol use behavior is mediated by the effect of olanzapine on cue-elicited craving. The final goal will be to examine whether genetic differences moderate the effects of olanzapine. [The polymorphism examined here involves the D4 dopamine receptor gene (DRD4), which has a variable number of tandem repeats (VNTR) in exon 3 (Van Tol et al., 1992). With respect to the DRD4 VNTR, individuals with at least one copy of an allele with 7 or more repeats are hereafter referred to as DRD4 L individuals, and individuals with alleles that have fewer than 7 repeats are hereafter referred to as DRD4 S individuals.]

In addition to laboratory studies on dopamine antagonists and alcohol craving (e.g., Modell et al., 1993; Hutchison et al., 2001), recent clinical reports have suggested that clozapine, a potent D4 receptor antagonist, reduces substance abuse among individuals with comorbid substance abuse/dependence (Green et al., 1999; Zimmet et al., 2000; Lee et al, 1998) and specifically, alcohol use (Drake et al., 2000). Animal studies have also suggested that clozapine reduces the voluntary intake of nicotine (Kameda et al., 2000). Given some of these early findings, we conducted a laboratory test of the effects of olanzapine on cue-elicited craving and craving after alcohol consumption among heavy social drinkers (Hutchison et al., 2001). We decided to test olanzapine because it also targets the D4 receptor, although not as strongly as clozapine, and because olanzapine had the best side effect profile among FDA approved medications that target dopamine receptors more broadly, and the D4 more specifically. This initial test demonstrated that olanzapine attenuated the effects of alcohol cues on two separate measures of urge to drink across two separate experimental sessions and that olanzapine prevented increases in urge to drink after alcohol consumption. With respect to the effects on urge to drink, the findings of this study are generally consistent with the theoretical premise that this appetitive behavior is partially mediated by mesolimbic dopamine activation.

To replicate and extend our previous results with olanzapine, a second study was designed to examine whether olanzapine (5 mg) reduced craving as compared to cyproheptadine (4 mg), which was used as an active control medication. It is important to note that there are no other published studies (to our knowledge) that have used such a stringent experimental control in a test of a pharmacological agent that targets alcohol craving in humans. For example, previous studies with naltrexone have utilized a placebo control only. The results from this investigation indicated that olanzapine and cyproheptadine produced equivalent levels of sedation. However, olanzapine significantly reduced craving before and after consuming alcohol, as compared to cyproheptadine (Hutchison et al., 2003). Moreover, there was a significant medication by DRD4 VNTR polymorphism interaction such that olanzapine reduced alcohol-elicited craving, particularly among DRD4 L individuals. To extend these findings, we conducted a 12 week, randomized, double-blind trial of olanzapine in the treatment of alcohol dependence (Hutchison et al., in press). Consistent with our previous studies, the results suggested that olanzapine reduced cue elicited craving and alcohol consumption significantly among DRD4 L individuals, but not DRD4 S individuals. Both of these last two studies were conducted at the Boulder GCRC.

Here, a double-blind, placebo-controlled 3 (Medication: olanzapine 5 mg, olanzapine 2.5 mg, vs. placebo) x 7 (Time: Baseline, 2, 4, 8, 12, 24, 36 weeks) mixed factorial design, where medication is a between-subjects factor and time is a within-subjects factor, will be used to test the treatment outcome hypotheses. Subjects will be randomly assigned to receive either olanzapine (5 mg), olanzapine (2.5 mg), or placebo for a period of 12 weeks such that there are equal numbers of DRD4 L individuals in each medication group. All subjects will also receive 7 sessions of medication management / supportive therapy (detailed below). Follow-up assessments will be obtained at 4, 8, 12 weeks (the end of treatment), 24 weeks, and 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 21-55 years of age with
* Alcohol Dependence

Exclusion Criteria:

* Medical Contraindications

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 304 (Actual)
Dates: Start 2002-09; Primary Completion 2010-05 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kent E Hutchison, Ph.D., Principal Investigator — The Mind Research Network
Locations (1):
- The Mind Research Network, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A double-blind, placebo-controlled 3 (Medication: olanzapine 5 mg, olanzapine 2.5 mg, vs. placebo) x 10 (Time: Baseline, 1, 2, 4, 6, 8, 10, 12, 24, 36 weeks). Subjects will be randomly assigned to receive either olanzapine (5 mg), olanzapine (2.5 mg), or placebo for a period of 12 weeks.
Pre-assignment Details: There is a discrepancy between number of participants enrolled, and number of participants started, due to some participants' ineligibility at screening. Therefore, the number enrolled refers to those participants who signed a consent form, whereas, the number started refers to those participants who were randomized to a treatment condition.
Groups:
- A - 2.5 mg Olanzapine: 2.5 mg Olanzapine
  olanzapine : 2.5 mg
- B - 5 mg Olanzapine: 5 mg Olanzapine
  olanzapine : 5 mg
- C - Placebo: placebo : placebo
Period: Overall Study
Arm/Group | A - 2.5 mg Olanzapine | B - 5 mg Olanzapine | C - Placebo
Started | 43 | 46 | 40
Completed | 14 | 21 | 13
Not Completed | 29 | 25 | 27
Not completed — Lost to Follow-up | 29 | 25 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A - 2.5 mg Olanzapine | B - 5 mg Olanzapine | C - Placebo | Total
Number analyzed (Participants) | 43 | 46 | 40 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 43 | 46 | 40 | 129
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 13 | 47
  Male | 26 | 29 | 27 | 82
Region of Enrollment [Number; unit: participants]
  United States | 43 | 46 | 40 | 129

OUTCOME MEASURES:

1. Primary Outcome: Drinks Per Drinking Day
Description: Drinks are measured as the number of standard alcoholic beverages consumed each day, assessed in varying lengths of time (i.e., 2 weeks, 4 weeks, 6 weeks, etc.). A standard alcoholic beverage is equivalent to: 1, 12 oz. regular beer; 1, 5 oz. glass of wine; 1, mixed drink with one1.5 oz shot; or 1, 1.5 oz shot. A drinking day is measured as any day of the week in which an alcoholic beverage is consumed. Data for drinks per drinking day is gathered using the "Time Line Follow Back" method in which participants are asked to recall their alcohol consumption day by day for a pre-defined set of time.
Time Frame: up to 36 weeks
Measure: Mean (Standard Deviation); unit: Drinks per drinking day
Arm/Group | A - 2.5 mg Olanzapine | B - 5 mg Olanzapine | C - Placebo
Number analyzed (Participants) | 43 | 46 | 40
Drinks per drinking day | 8.7 (5.3) | 8.9 (5.1) | 9.2 (5.4)

ADVERSE EVENTS:
Arm/Group | A - 2.5 mg Olanzapine | B - 5 mg Olanzapine | C - Placebo
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/46 | 0/40
Other Adverse Events (participants affected / at risk) | 2/43 | 2/46 | 0/40
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A - 2.5 mg Olanzapine (N=43) | B - 5 mg Olanzapine (N=46) | C - Placebo (N=40)
Diabetic Episode (General disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostasis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain/palpable mass (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No